CLINICAL TRIAL: NCT00406146
Title: Amodiaquine+Artesunate vs. Artemether-Lumefantrine for Uncomplicated Malaria in Ghanaian Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Ghana Medical School (Other)
Collaborators: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 91199 / 104. DAN.8-864; GHN-202-M03-M-00
Record Dates: First submitted 2006-11-13; First posted 2006-12-04 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2006-11

CONDITIONS: Uncomplicated Malaria
MeSH Terms: interventions — amodiaquine, artesunate drug combination; Artemether, Lumefantrine Drug Combination

INTERVENTIONS:
Drug: amodiaquine+artesunate/artemether-lumefantrine

SUMMARY:
Artemisinin combination therapies (ACT) are currently recommended for malaria treatment. Artemether-lumefantrine(A-L) and Artesunate+amodiaquine (A+A) have been the most commonly adopted of the recommended ACT regimens. In Ghana, A+A is the current first-line antimalarial treatment in Ghana, but there has been 1 efficacy report of this regimen in Ghana till date. Moreover, the safety of repeated treatments with ACT has been little studied. This study aims to evaluate the efficacy of A+A vs. A-L, as well as the safety of repeated treatments of these regimens in a longitudinal trial in which recruited children will be followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* microscopically confirmed acute uncomplicated falciparum malaria;
* temperature at screening 37.50C or more or history of fever 24 preceding enrollment;
* willingness to comply with follow up schedule;
* written informed consent by accompanying parent or guardian

Exclusion Criteria:

* features of severe malaria or danger signs of malaria
* known intolerance or allergy to any of the study medications
* known treatment with any of the study medications in the month preceding enrollment
* serious underlying disease that may mask outcome assessment

Ages: 6 Months to 14 Years | Sex: All
Age Groups: Child
Dates: Start 2004-10; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: George O. Adjei, MD, Principal Investigator — Dept. of Child Health, Korle Bu Teaching Hospital, Accra, Ghana; Bamenla Q. Goka, MBchB, Principal Investigator — Dept of Child Health, Korle Bu Teaching Hospital, Accra, Ghana; Jorgen A.L. Kurtzhals, MD, Ph.D, Principal Investigator — Dept. of Clinical Microbiology, Copenhagen University Hospital (Rigshospitalet), Copenhagen, Denmark
Locations (1):
- Korle Bu Teaching Hospital, Accra, Ghana

REFERENCES:
- [Derived] Adjei GO, Kurtzhals JA, Rodrigues OP, Alifrangis M, Hoegberg LC, Kitcher ED, Badoe EV, Lamptey R, Goka BQ. Amodiaquine-artesunate vs artemether-lumefantrine for uncomplicated malaria in Ghanaian children: a randomized efficacy and safety trial with one year follow-up. Malar J. 2008 Jul 11;7:127. doi: 10.1186/1475-2875-7-127. PMID 18620577